CLINICAL TRIAL: NCT05381896
Title: The Effect of Inspiratory Muscle Training on Postural Stability, Posture Perception and Trunk Rotation in Children With Adolescent Idiopathic Scoliosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Bezmialem Vakif University (Other); Istanbul Kent University (Other)
Responsible Party: Principal Investigator, Melih Zeren, asst. prof., Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bakircaymzeren06
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Adolescent Scoliosis
Keywords: postural stability; posture perception; inspiratory muscle training; adolescent idiopathic scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive conventional scoliosis exercise program for 1 hour, 6 days a week for 8 weeks. One exercise session will be supervised in a clinic per week, other sessions will be performed at home.
  Interventions: Other: Conventional Scoliosis Exercise Program
- Training Group (Experimental): In addition to the conventional scoliosis exercise program, patients in this group will also receive inspiratory muscle training for 15 minutes, twice a day, 6 days a week for 8 weeks. One exercise session will be supervised in a clinic per week, other sessions will be performed at home.
  Interventions: Other: Conventional Scoliosis Exercise Program; Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Conventional Scoliosis Exercise Program — Program will include breathing exercises, spinal stabilization and strengthening exercises, posture exercises and stretching execises.
Other: Inspiratory Muscle Training — Threshold IMT device will be used for the training. Training intensity will set at 30% of the maximum inspiratory pressure.
  Arms: Training Group

SUMMARY:
Trunk rotation and distortion of the rib cage, which are common in patients with adolescent idiopathic scoliosis, result in abnormal configuration of the diaphragm and intercostal muscles. This reduces the capacity of the respiratory muscles to produce force, and results in respiratory muscle weakness. The diaphragm, which is the major respiratory muscle, is also a component of the core muscles responsible for postural stability. Therefore, diaphragm muscle weakness results in deterioration of postural stability. Our aim in this study is to investigate the effect of inspiratory muscle training added to the routine scoliosis exercise program on postural stability and posture perception.

ELIGIBILITY:
Inclusion Criteria:

* Having adolescent idiopathic scoliosis with a Cobb angle of 20-50° diagnosed by an orthopedic surgeon

Exclusion Criteria:

* Having a documented diagnosis of neurological disorders
* Having a documented diagnosis of mental disorders which may affect cooperation
* Having a documented diagnosis of chronic airway diseases
* Having a documented diagnosis of orthopedic disorders which may affect mobility

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline postural stability test score in Biodex Balance System SD at 8 weeks | 8 weeks
Change from baseline limits of stability test score in Biodex Balance System SD at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Change from baseline "Walter Reed Visual Assessment Scale" at 8 weeks | 8 weeks
  Walter Reed Visual Assessment Scale evaluates posture perception. It consists of a visual test including seven items that deal with various aspects of the deformity. Each question has a set of five figures that represent degrees of severity of the deformity: spinal deformity, rib prominence, lumbar prominence, thoracic deformity, trunk imbalance, shoulder asymmetry and scapular asymmetry.
Change from baseline maximum inspiratory pressure (MIP) at 8 weeks | 8 weeks
Change from baseline maximum expiratory pressure (MEP) at 8 weeks | 8 weeks
Change from baseline angle of trunk rotation at 8 weeks. | 8 weeks
  Angle of trunk rotation will be evaluated using Bunnell scoliometer in forward bending position

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided